CLINICAL TRIAL: NCT01965054
Title: The Use of Fish Oil Supplementation in Treatment of Intrahepatic Cholestasis of Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics unresolved at the IRB at Elmhurst Hospital
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 12-1542
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Intrahepatic cholestasis of pregnancy; fish oil; omega-3; Docosahexaenoic acid,; eicosapentaenoic acid
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish Oil Supplement Group (Experimental): Receive the daily DHA pill and given a validated Itching Survey to assess maternal symptoms on admission and then weekly thereafter
  Interventions: Dietary Supplement: Fish Oil Supplement Group
- Control Group (No Intervention): Given a validated Itching Survey to assess maternal symptoms on admission and then weekly thereafter.

INTERVENTIONS:
Dietary Supplement: Fish Oil Supplement Group — 1 liquid gel pill (440mg omega-3 fatty acids from fish oil) taken daily, enrollment to delivery
  Other Names: DHA; Docosahexaenoic acid; Women's One A Day
  Arms: Fish Oil Supplement Group

SUMMARY:
Intrahepatic cholestasis of pregnancy (ICP) is a unique disease of the liver resulting in abnormal bile acid levels and liver function. The incidence of ICP ranges from 0.1 - 15.6%. Women diagnosed with ICP most often present with itching, which may be severe. More concerning, however, is the impact of ICP on adverse fetal and pregnancy outcomes, including preterm delivery, meconium exposure, fetal demise, and increased neonatal respiratory complications. The risk for fetal demise has been estimated to be 1-3%. The mechanism of fetal demise in ICP is unknown, and therefore cannot be reliably predicted. There is evidence to suggest that extremely elevated bile acids levels are associated with worse fetal outcomes, particularly levels greater than 40 μmol/L.

Ursodeoxycholic acid (UDCA) has anticholestatic effects, and is used to treat a variety of cholestatic liver diseases. Many studies have demonstrated superiority of UDCA over other agents, including dexamethasone and cholestyramine, for relief of maternal pruritus, improvement in transaminitis, reduction in serum bile acid concentrations, and improved pregnancy outcomes. As a result, UDCA is now widely used as first-line treatment for symptomatic relief in patients with ICP.

Docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) are two omega-3 long chain polyunsaturated fatty acids found in fish. DHA is known to play a key role in early fetal brain development, and has been associated with modest beneficial effects on neurodevelopmental and cognitive outcomes in children. In neonates with parental nutrition-induced cholestasis (PN-cholestasis), parental fish oil has been shown to be hepatoprotective not only for treatment of PN-cholestasis, but for prevention of cholestasis in premature infants at risk for the disease. Our hypothesis is that fish oil supplementation with DHA in women with ICP who are treated with UDCA will increase the rate of decline in serum total bile acid levels.

The incidence of ICP at a single hospital center in Queens, NY is estimated to be 5% secondary to a high concentration of patients from high-risk ethnic groups. High risk patients with bile acid levels greater than or equal to 40 μmol/L are managed aggressively with inpatient admission for continuous fetal monitoring, treatment with UDCA, and serial total bile acid levels weekly. These are patients are routinely offered early delivery after documented fetal lung maturity between 36 and 37 weeks gestation, or for any signs of fetal distress. This study is a prospective randomized controlled trial comparing weekly serum total bile acid levels in women admitted for inpatient management of ICP among women supplemented with a standard prenatal vitamin versus supplementation with a prenatal vitamin and DHA.

DETAILED DESCRIPTION:
Intrahepatic cholestasis of pregnancy (ICP) is a unique disease of the liver resulting in abnormal bile acid levels and liver function. In the literature, the incidence of ICP ranges from 0.1 - 15.6%.[1] Women diagnosed with ICP most often present with itching, which may be severe. More concerning, however, is the impact of ICP on adverse fetal and pregnancy outcomes, including preterm delivery, meconium exposure, fetal demise, and increased neonatal respiratory complications. The risk for fetal demise has been estimated to be 1-3%. The mechanism of fetal demise in ICP is unknown, and therefore cannot be reliably predicted. There is evidence to suggest that extremely elevated bile acids levels are associated with worse fetal outcomes, particularly levels greater than 40 μmol/L.[3] Ursodeoxycholic acid (UDCA) improves impaired hepatocellular secretion by stimulating canalicular bile acid transporter protein expression, and is now widely used as first-line treatment for symptomatic relief in patients with ICP. [1] Docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) are two omega-3 long chain polyunsaturated fatty acids found in fish. DHA is known to play a key role in early fetal brain development, and has been associated with modest beneficial effects on neurodevelopmental and cognitive outcomes in children.[2] In neonates with parental nutrition-induced cholestasis (PN-cholestasis), parental fish oil has been shown to be hepatoprotective not only for treatment of PN-cholestasis, but for prevention of cholestasis in premature infants at risk for the disease.[3-5] The incidence of ICP at a single hospital center in Queens, NY is estimated to be 5% secondary to a high concentration of patients from high-risk ethnic groups. High risk patients with bile acid levels greater than or equal to 40 μmol/L are managed aggressively with inpatient admission for continuous fetal monitoring, treatment with UDCA, and serial total bile acid levels weekly, and are routinely offered early delivery after documented fetal lung maturity between 36 and 37 weeks gestation, or for any signs of fetal distress. This study is a prospective randomized trial of women diagnosed with ICP prior to 36 weeks who are admitted to Elmhurst Hospital for inpatient observation. Women will be randomized to receiving a standard prenatal vitamin daily or a prenatal vitamin plus fish oil supplementation in addition to the standard UDCA 300mg by mouth three times daily. Dietary fish intake for each subject will be recorded. Total bile acid serum levels will be followed weekly, and fetal monitoring with daily non-stress tests will be performed on all women as per standard care for ICP at Elmhurst hospital. The primary outcome of interest is a 20% reduction in serum total bile acid levels in the treatment group compared to the control group at each time point. Secondary outcomes of interest include changes in maternal symptoms as measured using a validated itching score, changes in UDCA dosing, length of hospital stay, and neonatal outcomes including gestational age at delivery, Apgar scores, neonatal intensive care unit admissions, neonatal length of stay, meconium aspiration, birth weight, and perinatal mortality. Assuming 80% statistical power and a significance level of 0.05 to detect a 20% reduction in serum total bile acids in the treatment group compared to the placebo group, a total of 100 patients in each arm is needed.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women aged 18 years or older admitted to Elmhurst Hospital Center (EHC) for inpatient management of ICP due to a serum total bile acid level > 40 μmol/L, or serum total bile acid level > 10 μmol/L with elevated AST or ALT, are eligible for enrollment

Exclusion Criteria:

* Women < 18 years
* Women with allergies to fish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Bile acid levels | up to 9 months
  reduction in bile acid levels. Weekly (as part of standard hospital laboratory protocol for admission with intrahepatic cholestasis of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kohari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

REFERENCES:
- [Derived] Walker KF, Chappell LC, Hague WM, Middleton P, Thornton JG. Pharmacological interventions for treating intrahepatic cholestasis of pregnancy. Cochrane Database Syst Rev. 2020 Jul 27;7(7):CD000493. doi: 10.1002/14651858.CD000493.pub3. PMID 32716060